CLINICAL TRIAL: NCT03529955
Title: A Phase 2, Open Label Single Arm Study for Evaluating Safety & Efficacy of Apremilast in the Treatment of Cutaneous Disease in Patients With Recalcitrant Dermatomyositis
Brief Title: Evaluating Safety & Efficacy of Apremilast in the Treatment of Cutaneous Disease in Patients With Recalcitrant Dermatomyositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-978
Record Dates: First submitted 2018-04-24; First posted 2018-05-21 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Dermatomyositis, Adult Type
Keywords: dermatomyositis; apremilast; recalcitrant cutaneous disease
MeSH Terms: conditions — Dermatomyositis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dermatomyositis patients with refractory cutaneous disease (Experimental): Patients with dermatomyositis and refractory skin disease on steroids and one steroid-sparing agent.
  Interventions: Drug: Apremilast 30mg

INTERVENTIONS:
Drug: Apremilast 30mg — Patients with refractory cutaneous dermatomyositis will be started on apremilast 30 mg twice a day in addition to a stable dose of their treatment regimen (including steroids and steroid sparing agents).

SUMMARY:
With limited treatment options available for dermatomyositis, the investigators hypothesize that apremilast, a phosphodiesterase-4 (PDE-4) inhibitor, is a safe and efficacious add-on treatment in patients with refractory cutaneous dermatomyositis.

The study will investigate the efficacy, safety and toxicity of apremilast given at 30 mg twice daily to patients with refractory cutaneous dermatomyositis. Clinical response will be assessed at 1 and 3 months. Patients will also be evaluated for durability of their response for up to 6 months.

Treatment will be monitored with frequent clinical visits (0, 1, 3 and 6 months) and blood tests (CBC, CMP, creatine kinase, aldolase). Treatment will be discontinued at disease progression or unacceptable adverse events. Disease progression is defined as 4 points increase in the cutaneous dermatomyositis disease area and severity index (CDASI) score, worsening of muscle disease by manual muscle testing (MMT-8) score and 5 points increase in dermatomyositis life quality index (DLQI).

5 mm skin biopsies from lesional skin will be performed before treatment with apremilast and after 3 months of treatment for gene expression profiling and confirmatory immunohistochemical stains.

DETAILED DESCRIPTION:
1. Sponsor Name (PI): Carole Bitar, MD
2. Sub-PI: Erin Boh, MD, PhD; Brittany Stumpf, MD; Collaborator: Nakhle Saba, MD
3. # of Participants Sites: 1, Tulane University 4: Participant Countries: United States

II. PRODUCT INFORMATION

1. Study Title: A phase 2, open label single arm study for evaluating safety & efficacy of apremilast in the treatment of cutaneous disease in patients with recalcitrant dermatomyositis.
2. Clinical Phase: Phase II clinical trial
3. Primary Celgene Product: Apremilast

III. CONCEPT DESIGN AND RATIONAL

1. Therapeutic Area: Immunology
2. Specialty: Connective tissue disease
3. Disease State: Dermatomyositis

4-If other specify: None

5. Study Rationale: Dermatomyositis is an inflammatory disease that predominantly involves the skin with or without proximal muscle weakness. First line treatment for dermatomyositis is systemic steroids however due to long-term side effects, patients are usually treated with a steroid sparing agent. There is no known consensus on treatment guidelines for dermatomyositis and many anti- inflammatory medications have been successfully used. Tulane University is a referral center for recalcitrant dermatomyositis cases.The investigators present the case of a 57 y.o female patient with multidrug recalcitrant dermatomyositis showing complete remission of her skin disease with apremilast and improvement of her muscle disease. This patient was diagnosed with dermatomyositis. Over a 6-year period, she was treated with adequate trials of multiple immunosuppressive agents, including hydroxychloroquine, mycophenolate mofetil, azathioprine, methotrexate, soriatane, Intravenous immunoglobulin (IVIG), tacrolimus, chlorambucil, infliximab and rituximab. For the last four years, physicians were unable to lower corticosteroids below 40 mg per day. Her disease continued to flare despite these therapies. Chronic steroid use resulted in insulin dependent diabetes mellitus as well as other steroids associated side effects. While on stable doses of mycophenolate mofetil, prednisone and rituximab, the patient developed arthritis and was started on apremilast 30 mg twice a day. Two months into her treatment she noticed significant improvement of her skin disease and then nearly complete clearance of the skin. Her muscle weakness lagged behind and she noticed improvement after 9 months of being on apremilast with normalization of her aldolase and CK. The patient was able to wean off all immunosuppressive agents and prednisone. She was in remission for over 2 years and off all medications. She experienced a mild flare of skin disease recently and she resumed apremilast only and cleared immediately and continues on apremilast as a monotherapy. Patient experienced mild nausea and diarrhea with apremilast that improved four weeks into the treatment. She was able to discontinue insulin, lose weight and she has continued to be clear of both skin and muscle symptoms for over 1.5 years.

This case was accepted as a poster presentation at the 2018 Annual Meeting of the American Academy of Dermatology "Poster #: 6672 - Apremilast: a Potential Treatment for Dermatomyositis." Following this successful outcome, the investigators initiated apremilast in 3 other patients with recalcitrant dermatomyositis. Two patients had recalcitrant cutaneous disease and responded to add on therapy of apremilast in 2 months with significant improvement of their skin disease. The third patient had refractory dermatomyositis to several steroid-sparing agents and with severe muscle disease was started on apremilast for arthritis. She experienced significant improvement of her muscle weakness together with decrease in her muscle enzyme creatine kinase.

These very exciting findings triggered the idea of studying apremilast as an adjunct treatment for recalcitrant cutaneous disease in dermatomyositis patients. This is a novel idea; apremilast was never studied for dermatomyositis. Apremilast may have more advantages in dermatomyositis compared to other immunosuppressive treatments. Dermatomyositis patients may have lung involvement, and apremilast is an agent that doesn't have lung side effects in contrast to methotrexate for example which is one of the main steroid sparing agents used for dermatomyositis.

The pathogenesis of dermatomyositis is multifactorial with environmental, genetic and immune factors contribution.T helper-1 (Th1) and T helper-2 (Th2) immune pathways play a fundamental role in dermatomyositis.There is increase in proinflammatory cytokines including tumor necrosis factor alpha (TNF-α), interleukin (IL) 1, IL 6, and interferon (INF) α,γ shifting the immune balance to a Th1 response.Th1 immune response was also involved in the pathogenesis of interstitial pneumonia in the setting of dermatomyositis.IL4 released by lymphocytes infiltrating skin and muscles in dermatomyositis patients contributes to increase in Th2 response in conjunction with Th1 response.

Apremilast is a PD4-E inhibitor currently used for psoriasis and psoriatic arthritis.However, its usage on patients with dermatomyositis has not been investigated.

By inhibiting PDE-4 apremilast increases the level of cyclic adenosine monophosphate (c-AMP), leading to decreased expression of proinflammatory cytokines including TNF-α and INF-γ thus inhibiting Th1 response. Apremilast can also block Th2 response by interfering with the level of IL6 secreted by type2 macrophages.While the mechanism of action of apremilast in dermatomyositis is unknown, we suggest that apremilast can be a potential treatment option for dermatomyositis through interfering with Th1 and Th2 response.

Apremilast is a well-tolerated oral medicine with transient gastrointestinal side effects. Apremilast offers an additional treatment option for those patients with recalcitrant dermatomyositis, unresponsive to more conventional therapy.

6. Treatment and Dosing: Investigators will enroll patients seen at our facilities with a known diagnosis of dermatomyositis who are still experiencing cutaneous disease after a trial of systemic steroids and one steroid-sparing agent. Investigators will add apremilast to their treatment regimen according to the approved dosage for psoriasis and psoriatic arthritis: 10 mg orally one time on day 1, 10 mg orally twice daily on day 2, 10 mg orally in AM and 20 mg orally in PM on day 3, 20 mg orally twice daily on day 4, 20 mg orally in AM and 30 mg orally in PM on day 5, then 30 mg orally twice daily thereafter.

7. Brief Study Synopsis: With limited treatment options available for dermatomyositis, investigators hypothesize that apremilast, a phosphodiesterase-4 (PDE-4) inhibitor, is a safe and efficacious add-on treatment in patients with recalcitrant cutaneous dermatomyositis.

The study will investigate the efficacy, safety and toxicity of apremilast given at 30 mg twice daily to patients with recalcitrant cutaneous dermatomyositis. Clinical response will be assessed at 1 and 3 months. Patients will also be evaluated for durability of their response for up to 6 months.

Treatment will be monitored with frequent clinical visits (0, 1, 3 and 6 months) and blood tests (CBC, CMP, CK, aldolase). Treatment will be discontinued at disease progression or unacceptable adverse events. Disease progression is defined as a 4 points increase in CDASI score, worsening of muscle disease by MMT-8 score and 5 points increase in DLQI.

5 mm skin biopsies from lesional skin will be performed before treatment with apremilast and after 3 months of treatment for gene expression profiling and confirmatory immunohistochemical stains.

8. Sampling and correlative analysis

Although, the proposed mechanism of action of apremilast is though PDE-4 inhibition resulting in c-AMP upregulation, the exact biological process that leads to dermatological response in dermatomyositis remains ill-defined.Investigators propose to perform gene expression profiling (GEP) using RNA sequencing on skin biopsies collected before and after treatment with apremilast. In addition, we plan to confirm our GEP findings at the protein level using immunohistochemical (IHC) stains.

A. Tissue sampling and preparation

1. Tissue collection 5 mm punch biopsy from dermatomyositis skin lesions will be performed at baseline and another 5 mm punch biopsy will be performed at the 3-month time point. Each biopsy will be vertically split in two pieces and snap frozen on dry ice then it will be stored at -80C for further analysis with RNA sequencing and IHC stains.
2. RNA extraction At the end of all timeline collections, each skin biopsy will be mechanically broken down followed by mRNA extraction using the RNeasy extraction Kit from QIAGENzz. mRNA will then be stored at -80°C for subsequent RNA sequencing as detailed below.

B. Correlative Analysis

Determining the mechanism of action of apremilast in dermatomyositis.

1. Gene expression profiling RNA extracted form skin biopsies collected before and after in vivo treatment with apremilast (as detailed above) will be subjected to RNA sequencing. Illumina strand-specific TruSeq libraries will be prepared from the polyA selected RNA and subjected to 1x100 base sequencing on an Illumina HiSeq2500 machine. The number of samples proposed here (10 samples before treatment and 10 samples after treatment) is expected to yield sufficient statistical power for this approach; smaller numbers have been used in similar approaches to investigate drugs' mechanism of action (usually three samples).

   RNA-seq analysis will be performed in conjunction with the Tulane Cancer Crusaders Next Generation Sequence Analysis Core (Tulane Cancer Center - https://tulane.edu/som/cancer/research/core-facilities/cancer-crusaders/). Gene and isoform expression will be determined using RSEM and differential expression will be analyzed using EB-seq. Genes that are identified as differentially expressed between the two groups with a False Discovery Rate (FDR) of < 0.05 will be subjected to analysis by Ingenuity (IPA, Redwood City, CA). This analysis will group the identified genes into specific pathways, cell types, or disease process. A similar approach will be conducted using Gene Set Enrichment Analysis (GSEA). These experiments and GEP analysis will be performed in conjunction with our collaborator's (Dr. Nakhle Saba) lab, given his extensive experience in this field.
2. Protein analysis Information identified by Ingenuity or GSEA (signaling pathways, regulatory molecules, etc…) will be verified using IHC staining on select samples.

ELIGIBILITY:
Inclusion Criteria:

* Must understand the risks and the benefits/purpose of the study and provide signed and dated informed consent.
* Must be 18 years at time of signing the informed consent form.
* Willing to participate in all required evaluations and procedures in the study including the ability to swallow pills without difficulty.
* Patients must have a diagnosis of DM based upon the characteristic cutaneous findings proposed by Sontheimer[6] and/or a skin biopsy consistent with DM.
* Patients must be candidate for systemic therapy for their DM skin disease defined by inadequate response to aggressive sun protection along with the use of potent topical corticosteroids and/or immunomodulators.
* Patients with a diagnosis of dermatomyositis on steroid-sparing agent and/or systemic steroids (maximum dose of prednisone 1mg/Kg) and still having cutaneous disease activity of at least 5 on the CDASI scale.
* If on immunosuppressive treatments and/or steroids, patients must be on stable doses for at least 4 weeks (28 days).
* Patients must undergo age appropriate cancer screening.
* Females of childbearing potential (FCBP) must have a negative pregnancy test at screening (day 0 of the study and every month throughout the study). While on investigational product and for at least 28 days after taking the last dose of investigational product.

Exclusion Criteria:

* Increasing or changing dose of topical therapy within 14 days of study day 0 (including but not limited to topical corticosteroids, tacrolimus, pimecrolimus).
* Increasing or changing systemic steroids dosing within 28 days of study day 0.
* Increasing or changing dosing for concurrent therapy agents within 28 days or 5 half-lives of the biologic agent, whichever is longer, before study day 0: methotrexate, azathioprine, mycophenolate mofetil, hydroxychloroquine, dapsone, leflunomide, cyclosporine, biologic agents (anti-TNFs), IVIG, rituximab.
* History of any clinically significant (as determined by the investigators) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major uncontrolled disease.
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Pregnant or breastfeeding.
* Untreated Latent Mycobacterium tuberculosis infection or active tuberculosis infection as indicated by a positive Purified Protein Derivative (PPD) skin test or T-spot.
* Any condition, including the presence of laboratory abnormalities that places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Patients with acute dermatomyositis onset and rapid progression of muscle disease or significant systemic involvement including pulmonary diseases associated with DM.
* Prior major surgery or major life-threatening medical illness within 2 weeks.
* Inflammatory bowel disease, malabsorption or any other gastrointestinal motility disorders that limit the absorption of the study drug.
* Active hepatitis B or C infection with detectible viral nucleic acid in the blood or known Human Immunodeficiency Virus (HIV) positivity.
* Prior history of suicide attempt at any time in the patient's lifetime prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
* Active substance abuse or a history of substance abuse within 6 months prior to screening.
* Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
* Prior treatment with apremilast.
* Any severe systemic illness requiring IV antibiotics within the two weeks prior to initiation of the study drug.
* Malignancy or history of malignancy within the past four years, except for:

  * treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
  * treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 4 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Bitar, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and research resources generated by this study will be made available to the research community and to the public at large. This strategy includes, but not limited to, presentations (poster or oral) at local, national, and international meetings; published abstracts, and journal articles (peer reviewed). Contact information will be provided in publications for direct inquiries of researchers. Data generated from sequencing and gene expression profiling will be deposited into the Gene Expression Omnibus (GEO), NCBI, to be accessible by general public. The study protocol will be shared with other researchers on the clinical trial.gov website. No identified personal patient informations will be shared.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Thompson C, Piguet V, Choy E. The pathogenesis of dermatomyositis. Br J Dermatol. 2018 Dec;179(6):1256-1262. doi: 10.1111/bjd.15607. Epub 2017 May 24. PMID 28542733
- [Background] Giris M, Durmus H, Yetimler B, Tasli H, Parman Y, Tuzun E. Elevated IL-4 and IFN-gamma Levels in Muscle Tissue of Patients with Dermatomyositis. In Vivo. 2017 Jul-Aug;31(4):657-660. doi: 10.21873/invivo.11108. PMID 28652434
- [Background] Oda K, Kotani T, Takeuchi T, Ishida T, Shoda T, Isoda K, Yoshida S, Nishimura Y, Makino S. Chemokine profiles of interstitial pneumonia in patients with dermatomyositis: a case control study. Sci Rep. 2017 May 9;7(1):1635. doi: 10.1038/s41598-017-01685-5. PMID 28487565
- [Background] Maier C, Ramming A, Bergmann C, Weinkam R, Kittan N, Schett G, Distler JHW, Beyer C. Inhibition of phosphodiesterase 4 (PDE4) reduces dermal fibrosis by interfering with the release of interleukin-6 from M2 macrophages. Ann Rheum Dis. 2017 Jun;76(6):1133-1141. doi: 10.1136/annrheumdis-2016-210189. Epub 2017 Feb 16. PMID 28209630
- [Background] Hatemi G, Melikoglu M, Tunc R, Korkmaz C, Turgut Ozturk B, Mat C, Merkel PA, Calamia KT, Liu Z, Pineda L, Stevens RM, Yazici H, Yazici Y. Apremilast for Behcet's syndrome--a phase 2, placebo-controlled study. N Engl J Med. 2015 Apr 16;372(16):1510-8. doi: 10.1056/NEJMoa1408684. PMID 25875256
- [Background] Sontheimer RD. Dermatomyositis: an overview of recent progress with emphasis on dermatologic aspects. Dermatol Clin. 2002 Jul;20(3):387-408. doi: 10.1016/s0733-8635(02)00021-9. PMID 12170874
- [Background] Narla A, Dutt S, McAuley JR, Al-Shahrour F, Hurst S, McConkey M, Neuberg D, Ebert BL. Dexamethasone and lenalidomide have distinct functional effects on erythropoiesis. Blood. 2011 Aug 25;118(8):2296-304. doi: 10.1182/blood-2010-11-318543. Epub 2011 Apr 28. PMID 21527522
- [Background] Fiskus W, Saba N, Shen M, Ghias M, Liu J, Gupta SD, Chauhan L, Rao R, Gunewardena S, Schorno K, Austin CP, Maddocks K, Byrd J, Melnick A, Huang P, Wiestner A, Bhalla KN. Auranofin induces lethal oxidative and endoplasmic reticulum stress and exerts potent preclinical activity against chronic lymphocytic leukemia. Cancer Res. 2014 May 1;74(9):2520-32. doi: 10.1158/0008-5472.CAN-13-2033. Epub 2014 Mar 5. PMID 24599128
- [Background] Rosenwald A, Chuang EY, Davis RE, Wiestner A, Alizadeh AA, Arthur DC, Mitchell JB, Marti GE, Fowler DH, Wilson WH, Staudt LM. Fludarabine treatment of patients with chronic lymphocytic leukemia induces a p53-dependent gene expression response. Blood. 2004 Sep 1;104(5):1428-34. doi: 10.1182/blood-2003-09-3236. Epub 2004 May 11. PMID 15138159
- [Background] Li B, Dewey CN. RSEM: accurate transcript quantification from RNA-Seq data with or without a reference genome. BMC Bioinformatics. 2011 Aug 4;12:323. doi: 10.1186/1471-2105-12-323. PMID 21816040
- [Background] Leng N, Dawson JA, Thomson JA, Ruotti V, Rissman AI, Smits BM, Haag JD, Gould MN, Stewart RM, Kendziorski C. EBSeq: an empirical Bayes hierarchical model for inference in RNA-seq experiments. Bioinformatics. 2013 Apr 15;29(8):1035-43. doi: 10.1093/bioinformatics/btt087. Epub 2013 Feb 21. PMID 23428641
- [Background] Saba NS, Liu D, Herman SE, Underbayev C, Tian X, Behrend D, Weniger MA, Skarzynski M, Gyamfi J, Fontan L, Melnick A, Grant C, Roschewski M, Navarro A, Bea S, Pittaluga S, Dunleavy K, Wilson WH, Wiestner A. Pathogenic role of B-cell receptor signaling and canonical NF-kappaB activation in mantle cell lymphoma. Blood. 2016 Jul 7;128(1):82-92. doi: 10.1182/blood-2015-11-681460. Epub 2016 Apr 28. PMID 27127301
- [Background] Saba NS, Wong DH, Tanios G, Iyer JR, Lobelle-Rich P, Dadashian EL, Liu D, Fontan L, Flemington EK, Nichols CM, Underbayev C, Safah H, Melnick A, Wiestner A, Herman SEM. MALT1 Inhibition Is Efficacious in Both Naive and Ibrutinib-Resistant Chronic Lymphocytic Leukemia. Cancer Res. 2017 Dec 15;77(24):7038-7048. doi: 10.1158/0008-5472.CAN-17-2485. Epub 2017 Oct 9. PMID 28993409
- [Background] Akbulut S, Yilmaz M, Yilmaz S. Graft-versus-host disease after liver transplantation: a comprehensive literature review. World J Gastroenterol. 2012 Oct 7;18(37):5240-8. doi: 10.3748/wjg.v18.i37.5240. PMID 23066319
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Rider LG, Werth VP, Huber AM, Alexanderson H, Rao AP, Ruperto N, Herbelin L, Barohn R, Isenberg D, Miller FW. Measures of adult and juvenile dermatomyositis, polymyositis, and inclusion body myositis: Physician and Patient/Parent Global Activity, Manual Muscle Testing (MMT), Health Assessment Questionnaire (HAQ)/Childhood Health Assessment Questionnaire (C-HAQ), Childhood Myositis Assessment Scale (CMAS), Myositis Disease Activity Assessment Tool (MDAAT), Disease Activity Score (DAS), Short Form 36 (SF-36), Child Health Questionnaire (CHQ), physician global damage, Myositis Damage Index (MDI), Quantitative Muscle Testing (QMT), Myositis Functional Index-2 (FI-2), Myositis Activities Profile (MAP), Inclusion Body Myositis Functional Rating Scale (IBMFRS), Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI), Cutaneous Assessment Tool (CAT), Dermatomyositis Skin Severity Index (DSSI), Skindex, and Dermatology Life Quality Index (DLQI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S118-57. doi: 10.1002/acr.20532. No abstract available. PMID 22588740
- [Derived] Bitar C, Ninh T, Brag K, Foutouhi S, Radosta S, Meyers J, Baddoo M, Liu D, Stumpf B, Harms PW, Saba NS, Boh E. Apremilast in Recalcitrant Cutaneous Dermatomyositis: A Nonrandomized Controlled Trial. JAMA Dermatol. 2022 Dec 1;158(12):1357-1366. doi: 10.1001/jamadermatol.2022.3917. PMID 36197661

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 Patients were screened.
  39 Patients were excluded: 25 Patients didn't meet the inclusion criteria. 11 Patients were lost to follow up. 3 Patients had pregnancy plans.
Groups:
- Dermatomyositis Patients With Refractory Cutaneous Disease: Patients with dermatomyositis and refractory skin disease on steroids and one steroid-sparing agent.
  Apremilast 30mg: Patients with refractory cutaneous dermatomyositis were started on apremilast 30 mg twice a day in addition to a stable dose of their treatment regimen (including steroids and steroid sparing agents).
Period: Overall Study
Arm/Group | Dermatomyositis Patients With Refractory Cutaneous Disease
Started | 8
Completed | 6
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dermatomyositis Patients With Refractory Cutaneous Disease
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] | 54 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Cutaneous Disease Activity Severity Index (CDASI) [Mean (Standard Deviation); unit: units on a scale] — Cutaneous Disease Activity Severity Index (CDASI) This scale measures the cutaneous disease activity in dermatomyositis in 15 anatomical locations Scale: 0-100 0 indicates no activity 100 indicates maximum activity
  units on a scale | 29.8 (10.6)
Muscle Disease Activity Score (MMT-8) [Mean (Standard Deviation); unit: units on a scale] — Muscle Disease Activity Score (MMT-8) This scale measures the muscle disease in 8 anatomical locations Scale: 0-150 0 indicates severe disease 150 indicates full muscle activity
  units on a scale | 144.5 (6.9)
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: units on a scale] — Dermatology Life Quality Index (DLQI)
  This scale measures the impact of dermatological disease on quality of life Scale: 0-30 0 indicates no impairment of quality of life 30 indicates severe impairment of quality of life
  units on a scale | 15.1 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Analysis Would be Overall Response Rate Measured by the Number of Participants Experiencing at Least 4 Points Decrease in CDASI Activity Score at 3 Months.
Description: Cutaneous dermatomyositis disease area and severity index (CDASI) activity score is a validated tool to measure skin disease activity in dermatomyositis. The overall response rate (ORR) includes partial and complete responses. Complete response is defined by a CDASI activity score of zero. Partial response is defined by a decrease of CDASI activity score of at least 4 points. Calculation is performed as the CDASI activity score at 3 month(s) minus the score at baseline. Missing data will be handled using the last observation carried forward approach (LOCF).
  CDASI activity score: Units on a scale from 0-100. Higher scores represent worse outcome.
Time Frame: Data collected at 3 months after baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | Dermatomyositis Patients With Refractory Cutaneous Disease
Number analyzed (Participants) | 8
Participants | 7

2. Secondary Outcome: 2. The Secondary Endpoint Analysis Would be Safety as Measured by the Number of Participants Experiencing Adverse Events and Serious Adverse Events Occurring During 6 Months of Therapy and 1 Month Follow up.
Description: The proportion of participants experiencing adverse events and serious adverse events was measured over 7 months period (6 months during the study and 1 month follow up) using Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
  Grade refers to severity of the AE. The CTCAE displays Grades 1 to 5 with unique clinical descriptions of severity for each AE:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age- appropriate instrumental Activity of Daily Living (ADL) Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL Grade 4 Life-threatening consequences; urgent intervention indicated Grade 5 Death related to AE All adverse events subjects experienced were grade 1 or 2 which is mild to moderate in severity.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dermatomyositis Patients With Refractory Cutaneous Disease
Number analyzed (Participants) | 8
Participants
  Headache Grade 1-2 | 7
  Nausea Grade 1-2 | 5
  Diarrhea Grade 1-2 | 4
  Herpes Zoster Grade 1-2 | 2
  Influenza Grade 1-2 | 1
  Pneumonia Grade 1-2 | 1
  Acute sinusitis Grade 1-2 | 1
  Hypertension Grade 1-2 | 1
  Ocular pressure Grade 1-2 | 1

3. Secondary Outcome: An Additional Secondary Endpoint Analysis Would be Durability of Response Measured Participants CDASI Activity Score or Change in Their CDASI Activity Score at 6 Months Compared to 3 Months.
Description: The durability of response will be measured using the CDASI activity score at 6 months minus CDASI activity score at 3 months. Complete response durability is defined as zero or minus difference between CDASI activity score at 6 months and CDASI activity score at 3 months. Partial response durability is defined as >4 points difference between CDASI activity score at 6 months and CDASI activity score at 3 months. Missing data will be handled using the last observation carried forward approach (LOCF).
  CDASI activity score: Units on a scale from 0-100. Higher scores represent worse outcome.
Time Frame: Data collected at 6 months compared to data collected at 3 months
Population: 7 Patients were analyzed at 3 months mark, and 6 patients were analyzed at the 6 months mark.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CDASI Score at 3 Months; CDASI Score at 6 Months: Patients with dermatomyositis and refractory skin disease on steroids and one steroid-sparing agent.
  Apremilast 30mg: Patients with refractory cutaneous dermatomyositis were started on apremilast 30 mg twice a day in addition to a stable dose of their treatment regimen (including steroids and steroid sparing agents).
Arm/Group | CDASI Score at 3 Months | CDASI Score at 6 Months
Number analyzed (Participants) | 7 | 6
score on a scale | 16.9 (8.3) | 14 (6.4)

4. Secondary Outcome: An Additional Secondary Endpoint Analysis Would Assess Quality of Life as Measured at 3 Months Compared to Quality of Life Measured at 6 Months
Description: Dermatology Life Quality Index (DLQI) is a validated tool to measure quality of life in patients with skin disease. Complete response is defined by a DLQI of zero at 3, and 6 months. Partial response is defined by a decrease of DLQI of at least 5 points at 3, and 6 months compared to baseline. Calculation is performed as the DLQI at 3, and 6 months minus the score at baseline. Missing data will be handled using the last observation carried forward approach (LOCF).
  Units : Units on a scale from 0-30, higher scores represent worse outcome.
Time Frame: Data collected at 3 and 6 months after baseline visit
Population: 7 Patients were analyzed at 3 months mark, and 6 patients were analyzed at the 6 months mark.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DLQI Score at 3 Months; DLQI Score at 6 Months: Patients with dermatomyositis and refractory skin disease on steroids and one steroid-sparing agent.
  Apremilast 30mg: Patients with refractory cutaneous dermatomyositis were started on apremilast 30 mg twice a day in addition to a stable dose of their treatment regimen (including steroids and steroid sparing agents).
Arm/Group | DLQI Score at 3 Months | DLQI Score at 6 Months
Number analyzed (Participants) | 7 | 6
score on a scale | 6.3 (4.6) | 4.2 (2.1)

5. Other Pre Specified Outcome: An Additional Endpoint Analysis Would Assess the MMT-8 Score in Patients With Muscle Disease as Measured at 3 and 6 Months Compared to Baseline.
Description: MMT-8 (Manual Muscle Testing-8) score is a validated tool to assess muscle strength. Calculate the mean change in MMT-8 score at 3 and 6 month(s) compared to baseline in patients with muscle disease.
  Units: Units on a scale. Scale goes from 0-150. 150 is perfect strength.
Time Frame: Data collected at 3 and 6 months after baseline visit
Population: 7 Patients were analyzed at 3 months mark, and 6 patients were analyzed at the 6 months mark.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MMT-8 Score at 3 Months; MMT-8 Score at 6 Months: Patients with dermatomyositis and refractory skin disease on steroids and one steroid-sparing agent.
  Apremilast 30mg: Patients with refractory cutaneous dermatomyositis were started on apremilast 30 mg twice a day in addition to a stable dose of their treatment regimen (including steroids and steroid sparing agents).
Arm/Group | MMT-8 Score at 3 Months | MMT-8 Score at 6 Months
Number analyzed (Participants) | 7 | 6
score on a scale | 143.3 (10.9) | 144.5 (8.0)

6. Other Pre Specified Outcome: An Additional Endpoint is to Assess the Gene Expression Profiling and Immunohistochemistry Analysis Change on Skin Biopsies at 3 Months Compared to Baseline.
Description: Skin biopsies from lesional skin will be performed before treatment with apremilast and after 3 months of treatment to assess changes in gene expression profiling and immunohistochemistry stain. Gene expression profiling will be analyzed using inferential statistics with a False Discovery Rate (FDR) of < 0.05.
Time Frame: Data collected at 3 months after baseline visit
Measure: Number; unit: Change
Units Other Than Participants: Genes
Groups:
- Skin Biopsy at Baseline for Gene Expression Profiling; Skin Biopsy at 3 Months Into Apremilast Therapy for Gene Expression Profiling: Patients with dermatomyositis and refractory skin disease on steroids and one steroid-sparing agent.
  Apremilast 30mg: Patients with refractory cutaneous dermatomyositis were started on apremilast 30 mg twice a day in addition to a stable dose of their treatment regimen (including steroids and steroid sparing agents).
Arm/Group | Skin Biopsy at Baseline for Gene Expression Profiling | Skin Biopsy at 3 Months Into Apremilast Therapy for Gene Expression Profiling
Number analyzed (Participants) | 7 | 7
Number analyzed (Genes) | 39076 | 195
Change
  Down regulated genes | 0 | 123
  Up regulated genes | 0 | 72
Statistical Analysis 1: Comparison: Skin Biopsy at Baseline for Gene Expression Profiling vs Skin Biopsy at 3 Months Into Apremilast Therapy for Gene Expression Profiling; The student t test (paired) and ANOVA analysis of variance were used to assess the mean change in CDASI, MMT-8, DLQI and to compare the positive cell detection on immunohistochemistry for CCL5, pSTAT1 and pSTAT3 at baseline and 3 months post apremilast. All p values were two-sided, and values <0.05 were considered statistically significant. Analyses were performed using GraphPad Prism 8 (GraphPad Software Inc.). The last observation carried forward approach was used for missing values; Test type: Equivalence — The student t test (paired) and ANOVA analysis of variance were used to assess the mean change in CDASI, MMT-8, DLQI and to compare the positive cell detection on immunohistochemistry for CCL5, pSTAT1 and pSTAT3 at baseline and 3 months post apremilast. All p values were two-sided, and values <0.05 were considered statistically significant. Analyses were performed using GraphPad Prism 8 (GraphPad Software Inc.). The last observation carried forward approach was used for missing values; p = 0.01, ANOVA — The investigators hypothesized that genes identified as significantly differentially expressed between the two groups will have ≥2-fold change at p<0.01

7. Other Pre Specified Outcome: An Additional Endpoint is to Assess the Immunohistochemistry Analysis Change on Skin Biopsies at 3 Months Compared to Baseline.
Description: Skin biopsies from lesional skin will be performed before treatment with apremilast and after 3 months of treatment to assess changes in immunohistochemistry stain.
Time Frame: Data collected at 3 months after baseline visit
Population: 7 Skin biopsies were analyzed at baseline and at the 3 months mark. Changes in levels of activated (phosphorylated) STAT1 and STAT3 pre- and post-therapy were analyzed using immunohistochemistry. STAT 1 and STAT 3 measures were done on frozen sections using Positive Cell Detection analysis in QuPATH software. STAT 1 and STAT 3 were not measured in the blood, so the number represents the analysis performed in a QuPATH software representing the percentage of positive cell detection and H score.
Measure: Mean (Standard Deviation); unit: Percentage of positive cell detection
Groups:
- Skin Biopsy at Baseline for IHC; Skin Biopsy at 3 Months Into Apremilast Therapy for IHC: Patients with dermatomyositis and refractory skin disease on steroids and one steroid-sparing agent.
  Apremilast 30mg: Patients with refractory cutaneous dermatomyositis were started on apremilast 30 mg twice a day in addition to a stable dose of their treatment regimen (including steroids and steroid sparing agents).
Arm/Group | Skin Biopsy at Baseline for IHC | Skin Biopsy at 3 Months Into Apremilast Therapy for IHC
Number analyzed (Participants) | 7 | 7
Percentage of positive cell detection
  STAT1 | 96.2 (48.6) | 50.1 (28.6)
  STAT3 | 44.3 (25.3) | 17.4 (7.7)

ADVERSE EVENTS:
Time Frame: Over 6 months period.
Arm/Group | Dermatomyositis Patients With Refractory Cutaneous Disease
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dermatomyositis Patients With Refractory Cutaneous Disease (N=8)
Headache (Nervous system disorders) | 7 (7) — Grade 1-2
Nausea (Gastrointestinal disorders) | 5 (5) — Grade 1-2
Diarrhea (Gastrointestinal disorders) | 4 (4) — Grade 1-2
Herpes Zoster (Infections and infestations) | 2 (2) — Grade 1-2
Influenza (Infections and infestations) | 1 (1) — Grade 1-2
Pneumonia (Infections and infestations) | 1 (1) — Grade 1-2
Acute sinusitis (Infections and infestations) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) — Grade 1-2
Ocular pressure (Eye disorders) | 1 (1) — Grade 1-2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03529955/Prot_SAP_001.pdf